CLINICAL TRIAL: NCT04052568
Title: Effects of Psilocybin in Anorexia Nervosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00182516
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psilocybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental psilocybin (Experimental): Participants will have up to four doses of psilocybin.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will undergo up to four moderate to high dose psilocybin sessions. Dosing at the first session will be 20 mg. For subsequent sessions participants will either remain at their previous dose, or increase by increments of 5 mg up to a maximum of 30 mg.

SUMMARY:
This open-label pilot study seeks to investigate the safety and efficacy of psilocybin in persons with chronic anorexia nervosa (AN). Psilocybin has previously been demonstrated to decrease depression and anxiety and increase long-term positive behavior change in other populations. The investigators seek to determine whether similar changes can be safely produced in people with AN when psilocybin is administered in a supportive setting with close follow-up. The investigators' primary hypotheses are that psilocybin is safe to administer in people with AN, that it will reduce measures of anxiety and depression, and that it will lead to increased quality of life. The investigators will also assess a number of exploratory measures related to eating disorder pathophysiology.

ELIGIBILITY:
General Inclusion Criteria:

* Currently meet criteria for AN restricting subtype by Diagnostic and Statistical Manual 5th edition (DSM-5) criteria, and have a history of AN for at least 3 years prior to screening
* Have at least one prior attempt at treatment
* Be otherwise medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests (complete blood count, comprehensive metabolic panel, urine pregnancy test, urine toxicology screen).
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours of each drug administration. The exception is caffeine.

General Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of childbearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality, heart valve, or transient ischemic attack in the past year. Resting heart rate may be no less than 50 beats per minute unless cleared by a cardiologist.
* Epilepsy with history of seizures
* Type 1 diabetes
* First degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I Disorder
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) Score | 1 week post final psilocybin session
  The HADS is a 14-item self-report questionnaire that assesses both anxiety (7 questions) and depression (7 questions). Each question is scored on a 4-point Likert scale from 0-3, with higher scores indicating more severe symptoms.
Change in health related quality of life as assessed by the Eating Disorder Quality of Life Scale (EDQLS) | 2 months post final psilocybin session
  This is a 40-item self-report measure of health related quality of life that is specifically developed for eating disorder populations. Each question is rated on a 5 point scale from 1-5, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change in Eating Disorder Examination Questionnaire (EDE-Q) score | 1 month post final psilocybin session
  This is a 28-item self-report score that measures severity of eating disorder symptoms across four domains that each make up a sub-scale: dietary restraint, eating concern, weight concern, and shape concern. A global score is calculated by averaging sub-scale scores. Sub-scale and global scores range from 0-6 with higher scores indicating higher severity.
Change in Eating Disorder Examination (EDE) score | 1 month post final psilocybin session
  This is clinician-administered interview that measures severity of eating disorder symptoms across four domains that each make up a sub-scale: dietary restraint, eating concern, weight concern, and shape concern. A global score is calculated by averaging sub-scale scores.
Change in Body mass index (BMI) | 3 months post final psilocybin session
  This is a measure of body mass calculated from height and weight (Kg/m^2).
Change in Anorexia Nervosa Stages of Change Questionnaire (ANSOCQ) score | 1 month post final psilocybin session
  The ANSOCQ is a 20-item self-administered questionnaire that places respondents in one of the five stages of change based on Prochaska and DiClemente's model. The maximum raw score is 100, with higher scores indicating higher levels of motivation. An overall classification of the stage of change is obtained by dividing the raw score by 5.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Griffiths, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States